CLINICAL TRIAL: NCT07042256
Title: Feasibility of MR-Informed Adaptive Marker-less SBRT in Patients With Bilateral Hip Prostheses Undergoing SBRT for Localized Prostate Cancer
Acronym: HIP-PRO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAO-25-004; 2025-01091 (Other: Swissethics)
Record Dates: First submitted 2025-06-10; First posted 2025-06-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Localized Prostate Adenocarcinoma
Keywords: Bilateral hip prostheses; SBRT; Stereotactic body radiotherapy; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group study (Other): Assessment of low-field MR-informed adaptive marker-less SBRT for definitive treatment of localized prostate cancer in patients with bilateral hip prostheses.
  Interventions: Radiation: Low-field MR-informed adaptive marker-less SBRT for definitive treatment of localized prostate cancer in patients with bilateral hip prostheses

INTERVENTIONS:
Radiation: Low-field MR-informed adaptive marker-less SBRT for definitive treatment of localized prostate cancer in patients with bilateral hip prostheses — Low-field MR-informed adaptive marker-less SBRT

SUMMARY:
Hip replacements and prostate cancer are independently and both together increasing prevalent in the aging population. In the United States, the prevalence of hip prostheses among men was 1.1 million in 20101, with approximately 500,000 hip prostheses performed annually. Bilateral total hip replacement is recommended for patients with osteoarthritis affecting both hip joints. Approximately 10-25% of total hip replacement patients undergo bilateral procedures. Stereotactic body radiotherapy (SBRT) has been widely adopted as an effective treatment for localized prostate cancer, offering high precision and reduced treatment time due to conventionally fractionated radiotherapy without increasing toxicity or comprising oncological outcomes. Therefore, the use of SBRT for treatment of localized prostate cancer has significantly increased. A cohort study using data from 302 035 patients in the National Cancer Database showed that use of SBRT for prostate cancer increased from 0.2% in 2004 to 12.4% in 2020 in the United States.

However, both CT and MR-guided SBRT present unique challenges for patients with prostate cancer and bilateral hip prostheses. Metallic implants, such as hip prostheses, produce artifacts and magnetic susceptibility issues that can obscure MR imaging near the prosthetic sites, potentially complicating target contouring and planning. Given the close proximity of the prostate gland to the pelvis, which houses the hip joints, patients with bilateral hip prostheses may have significant imaging artifacts that could impair MR-guided radiotherapy quality. CT-based SBRT is less affected by metallic artifacts, but it lacks the soft-tissue resolution needed for precise prostate and OAR delineation, a gap MR imaging is uniquely positioned to fill.

Low-field MRI systems are less prone to susceptibility artifacts, including those originating from metallic implants. As a result, signal loss and distortion are expected to occur only in the immediate vicinity of the implant, making these systems particularly advantageous for imaging patients with hip implants. A prospective study quantitatively and qualitatively compared the magnitude of metal total hip arthroplasty-induced imaging artifacts in vivo between 1.5T (i.e. high-field) and 0.55T (low-field) MRI in 15 patients. Qualitative artifact magnitude was on average rated as moderate to small on 0.55T and as large to moderate on 1.5T by 2 fellowship-trained musculoskeletal radiologists. In addition, metal artifacts' areas and diameters were smaller on 0.55T when compared with 1.5T MRI for all sequences (each p>0.016).

Given the limitations of current imaging systems, the investigators propose a more flexible solution: a two-room system comprising a low-field MRI scanner for optimal image quality and a C-arm linear accelerator for rapid treatment delivery. Patient transfer between the MR device and the linear accelerator will be performed with a shuttle system which uses an air-bearing patient platform for both procedures. This setup would allow for high-quality imaging with reduced artifacts while ensuring efficient treatment times, addressing the current gap in SBRT for patients with bilateral hip prostheses. This shuttle system is MR-compatible and uses an air-bearing technology that allows the patient to be effortlessly moved by a transfer sled from MR scanner couch to linac without any movement on their part as it utilises the same patient platform with treatment using supports, immobilization devices and stereotactic tools for both procedures. This means that the patient is scanned and treated in the same position, minimising the risk of translational and/or rotational positional changes during transfer between both devices. Thus, maximum use of image-based planning data is possible. By integrating a low-field MRI scanner with a dedicated treatment delivery system, the investigators can overcome existing limitations and improve treatment precision for this growing patient population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of localized prostate cancer suitable for definitive SBRT based on a multidisciplinary tumour board recommendation and / or clinical practice guideline.
* Presence of bilateral hip prostheses labeled as MR safe or MR-conditional.
* ECOG performance status ≤ 2.
* Signed informed consent.
* Age ≥18 years -

Exclusion Criteria:

* Large body size that would not fit into the MRI-simulator bore
* Hip prosthesis that are labeled as MR unsafe;
* Contraindications to MRI including but not limited to:

  * Claustrophobia unmanageable by sedation
  * Electronic devices such as pacemakers, defibrillators, deep brain stimulators, cochlear implants that are labeled as MR unsafe, electronic devices labeled as MR safe or MR conditional are not a contraindication;
  * Metallic foreign body in the eye or aneurysm clips in the brain;
* Clinically significant concomitant diseases that would interfere with the study (e.g. hepatic dysfunction, cardiovascular disease).
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
MR-informed online adaptive definitive SBRT for localized prostate cancer | From enrollment to the end of treatment
  Evaluate the feasibility of MR-informed online adaptive definitive SBRT for localized prostate cancer using MR simulation and CBCT-based treatment delivery in patients with bilateral hip prostheses.

SECONDARY OUTCOMES:
Treatment toxicity | During treatment and up to 5 years after treatment, or death of the patient
  Treatment toxicity measured with Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Image quality | During treatment
  Difference in image quality and adapted contours as compared between 1.5 T and 0.55 T field strength MR scanners used for pre-treatment and intra-treatment simulation
Patient's wellbeing and comfort | During treatment
  Patients will be asked to report their comfort after simulation assessed with a 0 to 10 Numerical Rating Scale (NRS), with 0 representing complete absence of discomfort to 10 representing extreme discomfort.
Physicians decision certainty | During treatment
  Clinicians will be asked to report their clinical confidence with a 0 to 10 NRS, with 0 representing complete absence of clinical confidence to 10 representing extreme clinical confidence

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Guckenberger, Prof. Dr. med., Principal Investigator — University of Zurich

IPD SHARING:
Plan to Share IPD: No